CLINICAL TRIAL: NCT06010745
Title: A Randomized, Triple-blind, Placebo-controlled Study Evaluating the Efficacy of a Novel Dietary Ingredient for Improving Hair Growth and Skin's Appearance Among Healthy Adults
Brief Title: Effectiveness of a Novel Dietary Ingredient on Hair Growth and Skin's Appearance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nutrition 21, Inc. (Industry)
Collaborators: ALS Beauty and Personal Care (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALS 23-029
Record Dates: First submitted 2023-08-03; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Hair Thinning; Facial Skin Texture; Skin Ageing
Keywords: Hair Growth; Skin Texture
MeSH Terms: conditions — Alopecia | interventions — Biotin; Silicon

STUDY DESIGN:
Intervention Model Description: This is a six (6) month triple-blind, randomized, placebo-controlled study in women with self-perceived hair thinning/loss, with a six (6) month open-label arm in men using only the active product that will be conducted in parallel with the intervention study in women.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The primary intervention will utilize anonymized/coded products - anonymized/coded by the manufacturer and product codes only kept by supply chain and not directly maintained by study sponsor. The clinical test site will re-code the products, so the study will actually be triple-blind.
  Open-label products will be made with the active ingredients and this product will be labeled as an active - with no masking of identity to study sponsor, clinical site, or study participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active capsules (Active Comparator): Dietary ingredient standardized to deliver 10 mg of biotin and 10 mg of silicon per serving (1 capsule/serving).
  Interventions: Dietary Supplement: Biotin and silicon
- Placebo capsules (Placebo Comparator): The placebo comparator contains only inert ingredients (1 capsule/serving)
  Interventions: Dietary Supplement: Placebo
- open label (Other): Open-label arm that will involve men who only receive the active dietary ingredient capsules. This arm will run in parallel with the blinded study conducted in women.
  Interventions: Dietary Supplement: Biotin and silicon

INTERVENTIONS:
Dietary Supplement: Biotin and silicon — The active ingredient contains a standardized level of biotin (10 mg) and silicon (10 mg) per serving.
  Other Names: Lustriva
  Arms: Active capsules; open label
Dietary Supplement: Placebo — Inert ingredients only
  Arms: Placebo capsules

SUMMARY:
The objective of this study is to assess the effectiveness of a novel dietary ingredient containing biotin and silicon for promoting hair growth and improving skin's appearance with six months of continuous daily usage among healthy adults.

DETAILED DESCRIPTION:
Scientific problem:

Hair thinning and hair loss are problems that affect both men and women. A variety of diet, lifestyle, life-stage, ethnicity/race, and genetic factors contribute to the thinning and loss of hair. While hair loss is not a condition that is life-threatening, it is life-impacting. Hair loss negatively affects confidence and is associated with decline in quality of life While FDA-approved treatments do exist, access or ease of use may be difficult, or use limited to men. Ingredients like biotin, silicon, and herbals have been marketed for hair, skin, and nail benefits. The studies on their benefits are equivocal, requiring continued research investments to guide evidence-based recommendations for use. The availability of an oral supplement that is safe and effective for everyday use may present a new option for men and women concerned with hair thinning or hair loss.

Specific aims The objective of this randomized, triple-blind, placebo-controlled study is to assess the effectiveness of a novel dietary ingredient formulated with 10 mg of biotin and 10 mg of silicon for improving the appearance of hair and skin in a generally healthy adult population. The primary aim of this study will be to evaluate the impact of daily use on hair growth. In addition, the impact of supplementation on other hair and skin parameters will be evaluated. The study will include both analytical measures and a subjective questionnaire in order to connect analytical outcomes with observable changes in appearance.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with self-reported concerns with the appearance of their hair and/or skin (i.e., history of breaking hair / wrinkles or discoloration of the skin).
* In good general health as determined by ALS staff.
* Individuals who, at baseline, are free of any dermatological or systemic disorder, which would interfere with the results, at the discretion of the Investigator.
* Individuals who agree to provide a comprehensive medical history and concomitant medication list for review by ALS staff.
* Individuals who will read, understand and sign an informed consent document and photography release form.
* Individuals who agree to use the test product as instructed by the testing facility and complete the full course of the study.
* Individuals who agree to maintain a stable lifestyle with no significant changes in diet, supplements, medications, or exercise routine.
* Individuals who agree to maintain a consistent routine of washing their hair and skin.
* Individuals with natural hair only at start and for the duration of trial (no extensions, weaves, pieces, etc.). Dyed hair will be permitted for individuals who agree to maintain the same hair color for the study duration.
* Individuals who have not participated in another clinical study or for the past 30 days and agree to not concurrently participate in any other studies.
* Individuals who will agree to continue to use their current personal care products (e.g. shampoo, conditioner, hair spray, mousse, lotions, creams, sunscreen, cosmetics, etc.) for the duration of the study and agree to not incorporate any new products with the exception of those provided by ALS. Subjects must have a safe use history of their current products for at least 30 days prior to screening.
* Individuals who agree to maintain the same length, hair styling and coloring practices for the duration of the study.
* Individuals who agree not to utilize any new over the counter, commercial or other products that are marketed and promoted for enhancing aspects of their hair or skin (e.g., Viviscal®, BioSil®, Nutrafol®, etc.) for the entire duration of the study and confirms not using them one month prior to screening. This includes biotin-based supplements that provide 1000 micrograms or more biotin and/or contain biotin in combination with other ingredients promoted for hair and skin benefits.
* Individuals who agree to refrain from strenuous activity/exercise for at least 24 hours prior to each study visit.
* Individuals who agree to refrain from alcohol-containing food or beverages for at least 24 hours prior to each study visit.
* Individuals who agree to visit a 3rd party off-site laboratory and participate in a blood draw (N=40).
* Individuals who agree to avoid all tanning (sun or artificial such as tanning beds, sprays and other topical applications) and excessive sun exposure for the entire duration of the study and confirms avoiding these elements for 2 weeks prior to screening.

Exclusion Criteria:

* Individuals who have had a history of any acute or chronic disease that could interfere with or increase the risk on study participation.
* Individuals with an active (flaring) disease or chronic skin allergies (atopic dermatitis, eczema, psoriasis, severe acne), or had recently treated skin cancer (within the last 12 months) or currently undergoing treatment for cancer.
* Individuals with a history of drug or alcohol abuse in the 12 months prior to screening.
* Individuals with a history of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications (e.g., azathioprine, belimumab, cyclophosphamide, Enbrel, Imuran, Humira, mycophenolate mofetil, methotrexate, prednisone, Remicade, Stelara) and/or radiation as determined by study documentation.
* Individuals with damaged skin at or in close proximity to test sites (e.g., sunburn, tattoos, scars, excessive hair, or other disfigurations) that would impact study assessments.
* Individuals having severe hair loss or are completely bald.
* Individuals with white or very light-colored hair that is not able to be analyzed using the outlined instrumentation.
* Individuals who have any history, which, in the Investigator's opinion, indicates the potential for harm to the subject or could place the validity of the study in jeopardy.
* Individuals who have had any medical procedure, such as laser resurfacing, microdermabrasion, retinol or AHA treatments, hyaluronic injections, collagen, or chemical peels to the test sites within the last 6 months (including Botox, Restylyn, or other fillers).
* Individuals who are currently using or during the last 6 months have used, Retin A, or other Rx/OTC Retinyl A, or other astringent derived products or alpha hydroxyl acid treatments for photo-aging and fine lines/wrinkles.
* Individuals who have used any products or devices to promote scalp hair growth (e.g., finasteride, minoxidil, Rogaine, Propecia) within 6 months of screening; or refusal to refrain from any of these for the study duration.
* Individuals who have started, stopped, or changed hormone replacement therapy (HRT) within 6 months prior to screening.
* Subjects with history or presence of any clinically significant cardiovascular (light headedness/fainting or drops in blood pressure or recent myocardial infarction), respiratory (including uncontrolled asthma or allergies), renal, hepatic, gastrointestinal, hematologic, neurologic, any type of cancer that required radiation and/or chemotherapy for 1 year prior to study, metabolic disease or disorder, including guanidinoacetate methyltransferase deficiency and herpes (HSV-1), or any uncontrolled medical illness which in the opinion of the Investigator would jeopardize the safety of the subject, interfere with study assessments, or impact the validity of the study.
* Individuals who indicate that they are pregnant, planning a pregnancy or nursing.
* Individuals who have been medically diagnosed with Type I Diabetes.
* Individuals who have a known history of hypersensitivity to any cosmetics, personal care products, and/or fragrances.
* Individuals who are employees of the company.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Estimated)
Dates: Start 2023-08-11 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Hair growth and hair density | baseline, 3 months, 6 months
  Changes in the appearance of hair growth and hair thickness [bioinstrumental method; image analzysis using FotoFinder Medicam 1000]

SECONDARY OUTCOMES:
Appearance of global final lines and wrinkles | baseline, 3 months, 6 months
  Changes in the appearance of facial fine lines and wrinkles [assessed simultaneously using Canfield VISIA CR System; images evaluated using Vaestro Image Analysis Toolkit from Canfield]
Skin (facial) firmness | baseline, 3 months, 6 months
  Changes in firmness of facial skin [ Cutometer MPA 580] -measured in mm
Skin (facial) elasticity | baseline, 3 months, 6 months
  Changes in facial skin elasticity [Cutometer MPA 580] - measured in %
Skin hydration | baseline, 3 months, 6 months
  Changes in the water content of human skin [changes in skin conductance (AU-Arbitrary Units) using Corneometer CM 825]
Skin texture-Skin Smoothness | baseline, 3 months, 6 months
  Changes in skin texture [measured optically using VisioScan VC 98] - Evaluated using SELS (Surface Evaluation of the Living Skin)- SEsm index-AU- Arbitrary Units
Skin texture-Skin Roughness | baseline, 3 months, 6 months
  Changes in skin texture [measured optically using VisioScan VC 98] - Evaluated using SELS (Surface Evaluation of the Living Skin);- SEr index-AU- Arbitrary Units

OTHER OUTCOMES:
Self-Assessment Questionnaire | baseline, 3 months, 6 months
  Self-Assessment - Please answer the following questions by circling the response that best describes any changes you have noticed since starting this study (from +3 (greatly improved), +2 (moderately improved), +1 (slightly improved), 0 (no change), -1 (slightly worsened), -2 (moderately worsened), -3 (greatly worsened)
  1. Thickness of hair
  2. Overall hair growth
  3. Volume of hair
  4. Appearance of hair
  5. Hair breakage
  6. Hair quality
  7. Hair shine
  8. Hair strength
  9. Hair loss/shedding
  10. Scalp coverage
  11. Appearance of skin
  12. Skin tone
  13. Skin coloration
  14. Roughness of skin
  15. Skin elasticity
  16. Skin smoothness
  17. Facial wrinkles
  18. Facial fine lines
  19. Skin hydration
  20. Nail stregnth
  21. Nail breakage
  22. Nail growth
  23. Overall well-being
  24. Overall appearance
  Please provide any personal experience you want to share.
Plasma biotin status | baseline, 6 months
  Changes in plasma biotin status (ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan DeSantis, Principal Investigator — ALS Beauty and Personal Care
Locations (1):
- ALS Beauty and Personal Care, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalman, D. S., & Hewlings, S. J. (2021). A Randomized Double-Blind Evaluation of a Novel Biotin and Silicon Ingredient Complex on the Hair and Skin of Healthy Women. Journal of Clinical & Experimental Dermatology Research, 12(1), 1-5.